CLINICAL TRIAL: NCT01180777
Title: Dispensing Evaluation of Printed Etafilcon A With Polyvinylpyrrolidone (PVP) Contact Lenses
Brief Title: Dispensing Evaluation of Printed Etafilcon A With Polyvinylpyrrolidone (PVP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-1579AP
Record Dates: First submitted 2010-08-03; First posted 2010-08-12 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- etafilcon A (A)/etafilcon A (B)/etafilcon A (C) (Other): Printed etafilcon A Lens with PVP (A) worn first, then printed etafilcon A Lens with PVP (B) worn second, then printed etafilcon A Lens with PVP (C) worn the last. Each period consisted of approximately one week of daily lens wear.
  Interventions: Device: etafilcon A (A); Device: etafilcon A (B); Device: etafilcon A (C)
- etafilcon A (A)/etafilcon A (C)/etafilcon A (B) (Other): Printed etafilcon A Lens with PVP (A) worn first, then printed etafilcon A Lens with PVP (C) worn second, then printed etafilcon A Lens with PVP (B) worn the last. Each period consisted of approximately one week of daily lens wear.
  Interventions: Device: etafilcon A (A); Device: etafilcon A (B); Device: etafilcon A (C)
- etafilcon A (C)/etafilcon A (A)/etafilcon A (B) (Other): Printed etafilcon A Lens with PVP (A) worn first, then printed etafilcon A Lens with PVP (A) worn second, then printed etafilcon A Lens with PVP (B) worn the last. Each period consisted of approximately one week of daily lens wear.
  Interventions: Device: etafilcon A (A); Device: etafilcon A (B); Device: etafilcon A (C)
- etafilcon A (B)/etafilcon A (C)/etafilcon A (A) (Other): Printed etafilcon A Lens with PVP (B) worn first, then printed etafilcon A Lens with PVP (C) worn second, then printed etafilcon A Lens with PVP (A) worn the last. Each period consisted of approximately one week of daily lens wear.
  Interventions: Device: etafilcon A (A); Device: etafilcon A (B); Device: etafilcon A (C)
- etafilcon A (C)/etafilcon A (B)/etafilcon A (A) (Other): Printed etafilcon A Lens with PVP (C) worn first, then printed etafilcon A Lens with PVP (B) worn second, then printed etafilcon A Lens with PVP (A) worn the last. Each period consisted of approximately one week of daily lens wear.
  Interventions: Device: etafilcon A (A); Device: etafilcon A (B); Device: etafilcon A (C)
- etafilcon A (B)/etafilcon A (A)/etafilcon A (C) (Other): Printed etafilcon A Lens with PVP (C) worn first, then printed etafilcon A Lens with PVP (A) worn second, then printed etafilcon A Lens with PVP (C) worn the last. Each period consisted of approximately one week of daily lens wear.
  Interventions: Device: etafilcon A (A); Device: etafilcon A (B); Device: etafilcon A (C)

INTERVENTIONS:
Device: etafilcon A (A) — Daily wear contact lens
  Other Names: printed etafilcon A Lens with PVP (A)
Device: etafilcon A (B) — Daily wear contact lens
  Other Names: printed etafilcon A Lens PVP (B)
Device: etafilcon A (C) — Daily wear contact lens
  Other Names: printed etafilcon A Lens PVP (C)

SUMMARY:
The purpose of this study is to evaluate the lens fit (mechanical and cosmetic lens fit) of the printed etafilcon A with polyvinylpyrrolidone (PVP).

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be at least 18 years of age and less than 40 years of age.
2. The subject must be a light eye Caucasian female habitual soft contact lens wearer.
3. The subject must be concept acceptors for cosmetic and/or limbal ring lenses. A concept screening questionnaire will be used and top 3 box (in 5-point scale) is eligible.
4. The subject must have no known ocular or systemic allergies that might interfere with contact lens wear.
5. The subject must have no known systemic disease, or need for medication, which might interfere with contact lens wear.
6. The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and - 5.00D.
7. Any cylinder power must be ≤ -0.75D.
8. The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
9. The subject must have normal eyes (no ocular medications or ocular infection of any type).
10. The subject must read and sign the Statement of Informed Consent.
11. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

1. Ocular or systemic allergies or disease which might interfere with contact lens wear.
2. Systemic disease or use of medication which might interfere with contact lens wear.
3. Clinically significant (grade 3 or worse) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
4. Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
5. Any ocular infection.
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Any color deficiencies - to the best of the subject's knowledge.
8. Pregnancy or lactation.
9. Diabetes.
10. Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
11. Habitual contact lens type is toric, multifocal, or is worn as extended wear.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2010-08-01 (Actual); Study Completion 2010-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Cupertino, California
  - Los Angeles, California
  - San Jose, California
  - Jacksonville, Florida
  - Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an eight-site, randomized, 4-visit, bilateral crossover, dispensing trial.
Pre-assignment Details: Of those 95 enrolled subjects in this study, 3 did not meet the eligibility criteria, 6 prematurely discontinued from the study, and 6 excluded from the analysis due to protocol deviations.
Groups:
- All Subjects: All subjects who enrolled, randomized, and exposed to the study lenses. Subjects where randomized to a study arm and wore all three of the study lenses by study completion. Randomization was to the arms as outlined in the 'arms' section of the protocol.
Period: Overall Study
Arm/Group | All Subjects
Started | 92
Completed | 80
Not Completed | 12
Not completed — Protocol Violation | 6
Not completed — Poor lens fit | 4
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Subjects were to wear all three lenses over the course of the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 95
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 95

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit Acceptance
Description: Lens fit acceptance (whether acceptable or unacceptable) was assessed by the Investigator at dispensing.
Time Frame: 10-15 minutes post lens fit
Population: All subjects who successfully completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A (A) | Etafilcon A (B) | Etafilcon A (C)
Number analyzed (Participants) | 80 | 80 | 80
Number analyzed (Eyes) | 158 | 160 | 157
eyes
  Acceptable | 158 | 158 | 157
  Unacceptable | 0 | 2 | 0

2. Secondary Outcome: Binocular Snellen Visual Acuity (VA)
Description: Binocular Snellen VA was assessed at dispensing by Investigator using a Snellen vision chart. Subjects were analyzed based on their performance on a Snellen Vision chart exam in the study lenses in an effort to measure how well the lenses perform for vision correction.
Time Frame: 10-15 minutes post lens fit
Population: All subjects who successfully completed the study.
Measure: Number; unit: participants
Arm/Group | Etafilcon A (A) | Etafilcon A (B) | Etafilcon A (C)
Number analyzed (Participants) | 78 | 78 | 78
participants
  20/15 | 42 | 39 | 45
  20/20 | 36 | 39 | 33

3. Secondary Outcome: Corneal Staining
Description: Corneal staining type was graded in a 5-point scale over the 5 corneal regions by Investigator using a slit lamp; 0=none, 1=trace, 2=mild, 3=moderate, and 4=severe. Maximum grade of corneal staining type over the 5 corneal regions was categorized either absence or presence of corneal staining for the analysis.
Time Frame: After 6-9 days of lens wear
Population: All subjects who successfully completed the study.
Measure: Number; unit: eyes
Units Other Than Participants: eye
Arm/Group | Etafilcon A (A) | Etafilcon A (B) | Etafilcon A (C)
Number analyzed (Participants) | 80 | 80 | 80
Number analyzed (eye) | 160 | 154 | 158
eyes
  Central region grade > 0 | 4 | 6 | 3
  Inferior region grade > 0 | 34 | 25 | 44
  Nasal region grade > 0 | 2 | 6 | 7
  Superior region grade > 0 | 7 | 5 | 3
  Temporal region grade > 0 | 8 | 3 | 5

ADVERSE EVENTS:
Groups:
- All Subjects: Subjects were to wear all three lenses over the course of the study. Due to the non-ocular related AE, all subjects are summarized to report the occurrence of event.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 1/95
Other Adverse Events (participants affected / at risk) | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=95)
Appendicitis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires agreement and written authorization from the Sponsor